CLINICAL TRIAL: NCT05718804
Title: The Relationship Between Gut Microbiota and Sepsis-associated Acute Kidney Injury in Sepsis Patients：Multicenter Observational Study
Brief Title: Gut Microbiota and Sepsis-associated Acute Kidney Injury
Acronym: GMASAKI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Qinghai Provincial People 's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2022-016
Record Dates: First submitted 2023-01-10; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Sepsis; Acute Kidney Injury
Keywords: Sepsis-associated kidney injury; gut microbiota; metagenome; prognosis
MeSH Terms: conditions — Sepsis; Acute Kidney Injury | interventions — Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis-associated kidney injury: Sepsis patients and acute kidney injury No intervention
  Interventions: Other: Whether renal injury occurred and differences in intestinal flora
- Sepsis but no renal impairment: Sepsis patients without acute kidney injury
  Interventions: Other: Whether renal injury occurred and differences in intestinal flora

INTERVENTIONS:
Other: Whether renal injury occurred and differences in intestinal flora — Whether renal injury occurred and differences in intestinal flora
  Other Names: No intervention

SUMMARY:
Sepsis has emerged as one of the important life-threatening infectious diseases with high morbidity and mortality. Sepsis-associated kidney injury (SAKI) is one of the most common and serious complications of sepsis. It has been found that intestinal flora may affect the occurrence and development of a variety of diseases, and may also affect the pathogenesis of multiple SAKI, which is also regulated by host genetic factors. Therefore, the investigators speculate that gut microbiota composition may be associated with susceptibility to SAKI, and there are no studies reporting the association between gut microbiota and SAKI. The investigators intend to carry out a multicenter study in conjunction with the Department of Intensive Care of Qinghai Provincial People's Hospital. The structure and function of intestinal flora in septic patients with renal injury and septic patients less susceptible to renal injury are studied by 16S rDNA amplicon sequencing technology. The differences in composition, diversity and structural stability of intestinal flora between the two groups are analyzed to explore the genera that play a key role in the occurrence of the disease. By analyzing the differences between renal injury and inflammation levels in each group, the correlation between intestinal flora and SAKI, the possible influencing links involved, and the related factors affecting the prognosis of SAKI were revealed. The results of this study are helpful to further elucidate the pathogenesis of SAKI and provide new ideas and methods for the prevention and treatment of SAKI.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years；Meet the sepsis definition and diagnostic criteria of Sepsis-3.0 guidelines；No previous history of hypertension or diabetes; No underlying kidney disease such as nephrotic syndrome, no history of rheumatic immune system disease; Normal renal function before onset.

Exclusion Criteria:

* Patients with hypertension, diabetes, coronary heart disease, tumor, rheumatism immune system disease and other related diseases that may cause kidney injury; Patients with abnormal renal function before onset; Patients with nephrotic syndrome and other underlying kidney disease; Long-term oral administration of drugs with kidney injury; Previous history of gastrointestinal surgery; No diarrhea related diseases or other gastrointestinal diseases in the past 1 month; The use of antibiotics and probiotics in the past 1 month; Exclusion of other primary or secondary renal damage factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sepsis patients who met the inclusion criteria were admitted to the First Affiliated Hospital of Xi'an Jiaotong University and Qinghai Provincial People 's Hospital during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in gut microbiota composition between the two groups | Within 24 hours of patient enrollment
  The differences in the composition of intestinal flora between the two groups were analyzed to identify the correlation with AKI

SECONDARY OUTCOMES:
IL-6 | Within 24 hours of patient enrollment
  the concentration of Interleukin 6 (IL-6)

CONTACTS AND LOCATIONS:
Locations (1):
- First affliated hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No